CLINICAL TRIAL: NCT04320186
Title: Community Influences Transitions in Youth Health II - Center for the Study of Community Health
Brief Title: Community Influences Transitions in Youth Health (CITY) Health II - Center for the Study of Community Health
Acronym: CH-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Davies, Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150219009
Record Dates: First submitted 2020-03-06; First posted 2020-03-24 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Sexually Transmitted Diseases; HIV Infections
Keywords: prevention and control; young adults; african americans; education entertainment; condom use
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: two groups design with approximately equal allocation, but assignment based on respondent drive sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Participants viewed informational video content plus entertainment content
  Interventions: Behavioral: Entertainment education; Other: video
- Control (Placebo Comparator): Participants viewed entertainment content only
  Interventions: Behavioral: Entertainment education

INTERVENTIONS:
Behavioral: Entertainment education
Other: video — video
  Arms: Treatment

SUMMARY:
The purpose of this protocol is to develop and evaluate an HIV prevention Entertainment Education (EE) intervention aimed at reaching underserved, at-risk African Americans, aged 18-25 years, living in disadvantaged urban neighborhoods in the Birmingham area.

DETAILED DESCRIPTION:
The goal of this 5 year project is to promote HIV testing and improve HIV-related risk behaviors (e.g. condom use, substance use before sex, regular Sexually Transmitted Infection (STI) testing) via population-sensitive and population-specific HIV prevention videos that are appealing, evidence-based, scalable, and sustainable to the target population. Formative research was conducted in Phase I (Year 1-2), to pre-test the questionnaire and gather in-depth data (via focus groups, intercept interviews, and individual structured interviews) to inform intervention development. Phase 2 of the project involved developing, delivering, and subsequently evaluating the efficacy of peer-driven EE HIV prevention messaging to broader social networks via a social media platform, with the platform contingent on formative data. An HIV education video series, "The Beat HIVe", was produced and served as intervention materials for the quasi-experimental research project. Respondent Driven Sampling (RDS) was used to access and use the social networks of high-risk youths as channel and agents for change. RDS is a recent innovative adaptation of chain-referral network sampling that provides peer-driven access to hard-to-reach subpopulations while reducing sampling biases associated with conventional snowball sampling.

ELIGIBILITY:
Inclusion Criteria:

African American young adults Aged 18-25 Living in the Birmingham USA Competent to give informed consent

Exclusion Criteria:

Obvious psychosis, dementia, inability to hear. Plan to move within the next 6 months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 334 (Actual)
Dates: Start 2015-04-03 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
HIV Knowledge Questionnaire-18 | Baseline
  This scale assess an individual level of HIV-related knowledge. For each of the 18 true/false, HIV- related questions, a score of 1 was assigned to each 'correct' answer. Assessments were based on the analysis of the summation of these scores, which had a possible range of 0 to 18, whereby higher scores indicated greater knowledge of HIV.
HIV Knowledge Questionnaire-18 | 3 months
  This scale assess an individual level of HIV-related knowledge. For each of the 18 true/false, HIV- related questions, a score of 1 was assigned to each 'correct' answer. Assessments were based on the analysis of the summation of these scores, which had a possible range of 0 to 18, whereby higher scores indicated greater knowledge of HIV.
HIV Knowledge Questionnaire-18 | 6 months
  This scale assess an individual level of HIV-related knowledge. For each of the 18 true/false, HIV- related questions, a score of 1 was assigned to each 'correct' answer. Assessments were based on the analysis of the summation of these scores, which had a possible range of 0 to 18, whereby higher scores indicated greater knowledge of HIV.
Perceived HIV-related Stigma | Baseline
  The scores are scaled in the positive direction implying that the higher the score, the higher the level of stigma. The possible overall stigma score ranges from 40 to 160, low-level stigma is between 25th percentile and 50th percentile (40-80), middle-level stigma is between 50th percentile and 75th percentile (81-120), while high-level stigma is for values greater than 75th percentile (121-160).
Perceived HIV-related Stigma | 3 months
  The scores are scaled in the positive direction implying that the higher the score, the higher the level of stigma. The possible overall stigma score ranges from 40 to 160, low-level stigma is between 25th percentile and 50th percentile (40-80), middle-level stigma is between 50th percentile and 75th percentile (81-120), while high-level stigma is for values greater than 75th percentile (121-160).
Perceived HIV-related Stigma | 6 months
  The scores are scaled in the positive direction implying that the higher the score, the higher the level of stigma. The possible overall stigma score ranges from 40 to 160, low-level stigma is between 25th percentile and 50th percentile (40-80), middle-level stigma is between 50th percentile and 75th percentile (81-120), while high-level stigma is for values greater than 75th percentile (121-160).
Condom Use Self-Efficacy Scale | Baseline, 3- and 6 months
  This is a 28 item self-report questionnaire which elicits responses using a five-point Likert scale format, ranging from 'strongly disagree' to 'strongly agree'. Each of the responses is scored as follows: 'strongly disagree' = 0, 'disagree' = 1, 'undecided' = 2, 'agree' = 3 and 'strongly agree' = 4. After reversing for negatively worded items, scores are summed. The possible range of scores is 0-112, with higher scores indicating greater condom use self-efficacy.
Condom Use Self-Efficacy Scale | Baseline
  This is a 28 item self-report questionnaire which elicits responses using a five-point Likert scale format, ranging from 'strongly disagree' to 'strongly agree'. Each of the responses is scored as follows: 'strongly disagree' = 0, 'disagree' = 1, 'undecided' = 2, 'agree' = 3 and 'strongly agree' = 4. After reversing for negatively worded items, scores are summed. The possible range of scores is 0-112, with higher scores indicating greater condom use self-efficacy.
Condom Use Self-Efficacy Scale | 3 months
  This is a 28 item self-report questionnaire which elicits responses using a five-point Likert scale format, ranging from 'strongly disagree' to 'strongly agree'. Each of the responses is scored as follows: 'strongly disagree' = 0, 'disagree' = 1, 'undecided' = 2, 'agree' = 3 and 'strongly agree' = 4. After reversing for negatively worded items, scores are summed. The possible range of scores is 0-112, with higher scores indicating greater condom use self-efficacy.

SECONDARY OUTCOMES:
Timeline Followback | 6 months
  Assesses sexual activity over the previous 90-days. The baseline assessment collected sexual risk behavior data for the 3 months prior to enrolling in the study; the 3-month data collection visit examined participant's sexual risk behavior in the 90 days since their baseline visit; and their 6-month data collection visit used TLFB to record sexual risk behavior since their last visit. Following each interview, TLFB data are coded in accordance with a discrete coding algorithm that allows the research team to summarize all of this information directly on the daily blocks on the calendar.
HIV Testing Questionnaire | 6 months
  HIV testing uptake-after initial education. Participants were asked if they wanted to take a free and optional HIV test. If the participant declined they were asked additional 6 questions about their reason for declining. If they accepted the HIV test, they were asked additional 20 questions regarding how often they tested, knowledge of testing resources, sexual practices, and reason for accepting a test. This questionnaire was developed by study staff and is not scored.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Davies, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davies SL, Smith TL, Murphy B, Crawford MS, Kaiser KA, Clay OJ. CITY Health II - using entertainment education and social media to reduce HIV among emerging adults: A protocol paper for the Beat HIVe project. Contemp Clin Trials. 2020 Dec;99:106167. doi: 10.1016/j.cct.2020.106167. Epub 2020 Oct 5. PMID 33031956